CLINICAL TRIAL: NCT00448422
Title: A Multicenter, Double-Blind, Randomized Study to Compare the Safety and Efficacy of Prulifloxacin Versus Placebo in the Treatment of Acute Gastroenteritis in Adult Travelers
Brief Title: Safety and Efficacy of Prulifloxacin vs Placebo in Treatment of Acute Gastroenteritis in Adult Travelers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Optimer Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Y.K. Shue, Optimer Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPT-099-002
Record Dates: First submitted 2007-03-15; First posted 2007-03-16 (Estimated); Last update posted 2010-09-27 (Estimated); Status verified 2010-09

CONDITIONS: Acute Bacterial Gastroenteritis
Keywords: Traveler's; Diarrhea
MeSH Terms: conditions — Diarrhea | interventions — prulifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Tablet
  Interventions: Drug: prulifloxacin
- 2 (Placebo Comparator): Tablet
  Interventions: Drug: prulifloxacin

INTERVENTIONS:
Drug: prulifloxacin — Tablet

SUMMARY:
The objective of this pivotal Phase III study is to investigate the safety and efficacy of prulifloxacin versus placebo in the treatment of patients with acute bacterial gastroenteritis (traveler's diarrhea.

DETAILED DESCRIPTION:
This double-blind trial will compare the safety and efficacy of prulifloxacin versus placebo in adult travelers with acute gastroenteritis characterized by diarrhea with one or more of the following signs or symptoms: nausea, vomiting, abdominal pain or cramping, fecal urgency, moderate to severe other gastrointestinal-related symptoms, or tenesmus of <72 hours duration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute bacterial gastroenteritis
* Traveler from an industrialized country
* Capable of giving Informed Consent

Exclusion Criteria:

* Fever (>100.3 degrees)
* Pregnant or Breast Feeding or Not using adequate birth control
* Known or Suspected (co-)Infection with non-bacterial pathogen
* Symptoms of acute gastroenteritis of >72 hours duration
* Bloody Diarrhea
* Concomitant antibacterial with activity against enteric bacterial pathogens
* History of IBD
* Unable/Unwilling to comply with study protocol
* Greater than two doses of an antidiarrheal medication within 24 hours
* > 2 doses of anti-diarrheal medication within 24 hours
* Antimicrobial treatment within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2006-12; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Time to Last Unformed Stool (TLUS) | End of Therapy

SECONDARY OUTCOMES:
Microbiologic eradication rates | End of therapy/study
Clinical cure based on relief of signs and symptoms | End of therapy/study

CONTACTS AND LOCATIONS:
Overall Officials: Robert Steffen, MD, Study Director — University of Zurich
Locations (1):
- Goa Medical College, Bambolim, Goa, India